CLINICAL TRIAL: NCT06809322
Title: Vorasidenib as Maintenance Treatment After First-line Chemoradiotherapy in IDH-mutant Grade 2 or 3 Astrocytoma: a Placebo-controlled, Triple-blind, Randomized Phase III Study (VIGOR)
Brief Title: Vorasidenib Maintenance for IDH Mutant Astrocytoma
Acronym: VIGOR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Canadian Cancer Trials Group (Network); Olivia Newton-John Cancer Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EORTC -2427-BTG; 2024-519404-27-00 (EU CTIS Number); CE.10 (Other: Canadian Cancer Trials Group (CCTG))
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: IDH-mutant Grade 2 or 3 Astrocytoma
Keywords: Astrocytoma; IDH-mutant grade 2 or 3; Vorasidenib; Placebo- controlled; Triple-blinded; Phase III study
MeSH Terms: conditions — Astrocytoma | interventions — vorasidenib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Participants will receive vorasidenib orally once daily at a dose of 40 mg in continuous 28-day cycles up to 5 years or until disease progression, unacceptable toxicity, or withdrawal of patient consent.
  Interventions: Drug: Vorasidenib
- Control arm (Placebo Comparator): Participants will receive a matched oral vorasidenib placebo once daily in continuous 28-day cycles until disease progression, unacceptable toxicity, or withdrawal of patient consent for up to 5 years.
  Interventions: Drug: Vorasidenib Placebo

INTERVENTIONS:
Drug: Vorasidenib — Vorasidinib will be administered orally once daily at a dose of 40 mg in continuous 28-day cycles
  Arms: Experimental arm
Drug: Vorasidenib Placebo — Matched oral vorasidenib placebo will be administered once daily in continuous 28-day cycles
  Arms: Control arm

SUMMARY:
The main goal of VIGOR is to demonstrate that vorasidenib maintenance therapy improves locally assessed progression-free survival (PFS) from enrolment compared to placebo in patients with IDH-mutant, CNS5 WHO Grade 2 or 3 astrocytoma following the completion of first-line chemoradiotherapy.

The primary endpoint is Progression-free survival (PFS), as assessed locally from the date of enrolment using the RANO 2.0 criteria.

In this a comparative, randomized (1:1), triple blinded, multicentre phase III superiority trial with one stopping rule for efficacy and futility after end of enrolment, participants in the experimental arm will receive vorasidenib orally once daily at a dose of 40 mg in continuous 28-day cycles while participants in the control arm will receive a matched oral placebo once daily in continuous 28-day cycles

DETAILED DESCRIPTION:
Diffuse gliomas are the most common primary brain tumors in adults and are associated with high morbidity and mortality. Approximately 25% of diffuse gliomas harbour mutations in the isocitrate dehydrogenase (IDH) 1 or 2 genes. Among IDH-mutated gliomas, IDH-mutant astrocytoma is the most common diagnosis and occurs mainly in adults in their thirties or forties. Most cases correspond to CNS5 WHO grade 2 and 3, while grade 4 tumors are rare. The prognosis of grade 2 and 3 tumors is significantly better (median overall survival times up to 10 years) than that of grade 4 tumors (median overall survival times around 3-7 years).

According to international guidelines and based on randomized clinical trials, treatment options for IDH-mutated astrocytoma after maximum safe neurosurgical resection include active surveillance or radiotherapy followed by chemotherapy with procarbazine, lomustine and vincristine (PCV) or temozolomide. An active surveillance strategy, however, can be recommended for patients with oligodendroglioma grade 2 or astrocytoma grade 2 with particularly favourable prognostic factors, such as absence of neurological deficits and limited tumor burden. Despite this multimodal treatment, IDH-mutant astrocytomas recur and ultimately lead to patient death, with median progression-free survival times around 7 years and overall survival times of approximately 9-11 years. Novel treatment strategies are needed to extend the survival of these patients.

Recently, the international randomized placebo-controlled phase III INDIGO trial has shown considerable efficacy on progression free survival of the mutant IDH inhibitor vorasidenib in patients with IDH-mutant diffuse grade 2 gliomas that were considered candidates for an active surveillance strategy by the treating physician. Vorasidenib (AG881) is an orally available brain-penetrant dual inhibitor of mutant IDH1 and IDH2 proteins. INDIGO enrolled patients with residual or recurrent non-enhancing grade 2 IDH-mutant glioma who had not received prior radiotherapy or chemotherapy. Participants received either vorasidenib (40 mg once daily) or a matched placebo, given continuously in 28-day cycles. From January 2020 through February 2022, a total of 331 participants were randomly assigned to receive vorasidenib (168 participants) or placebo (163 participants ). The image-based progression-free survival was significantly longer for participants in the vorasidenib group than in the placebo group: 27.7 months (95% CI, 17.0 to non-estimable) vs 11.1 months (95% CI, 11.0-13.7), with a hazard-ratio for disease progression or death of 0.39 (95% CI, 0.27-0.56, p<0.001). Additionally, time to next intervention was significantly delayed in the vorasidenib group as compared to the placebo group with a hazard ratio of 0.26 (95% CI, 0.15-0.43, p<0.001). Adverse events leading to treatment interruption occurred in 3.6% of the vorasidenib group and 1.2% of the placebo group. An increased alanine amino transferase level of grade 3 or higher occurred in 9.6% of participants receiving vorasidenib and in none of the participants receiving placebo. Overall, based on the INDIGO trial data, registrational approval by the FDA was granted in August 2024 and EMA approval is expected. Vorasidenib is likely to enter routine clinical practice for patients with IDH-mutant gliomas that do not require immediate chemoradiotherapy.

In the current trial, the investigator will evaluate whether adding vorasidenib as maintenance therapy after completion of standard chemoradiotherapy in patients with astrocytoma, IDH-mutant, CNS5 WHO Grade 2 or 3 prolongs progression-free survival compared to placebo. This trial will also explore the effect of vorasidenib maintenance treatment on overall survival, response rate, time to next intervention, toxicity, health-related quality of life, neurological symptoms, and neurocognitive function. Additionally, this trial will enable translational research through the analysis of tissue samples, liquid biopsies (blood samples), and neuroimaging data.

Overall, VIGOR aims to establish a new standard of care for IDH-mutated, CNS5 WHO Grade 2 or 3 astrocytoma by incorporating maintenance targeted therapy with vorasidenib into the current standard of care chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Before participant's enrolment, written informed consent must be given according to ICH/GCP, and national/local regulations.
* Age ≥ 18 years
* Integrated diagnosis of astrocytoma, IDH-mutant, WHO CNS5 grade 2 or 3, per local assessment
* Documented IDH1 or IDH2 mutation based on local testing of tumour tissue
* At least 1 prior surgery for glioma (biopsy, partial resection, gross-total resection)
* Completed first-line standard of care radiotherapy (minimum 50.4 Gy, photons or protons allowed) followed by SoC adjuvant chemotherapy (i.e., either 4-12 cycles of temozolomide or 2-6 cycles of PCV).
* Adequate bone marrow function: absolute neutrophil counts ≥ 1.5 x 109/L, haemoglobin ≥ 9 g/dL, platelets 100 x 109/ L.
* Adequate renal function: serum creatinine ≤ 2.0 x ULN, or creatine clearance > 40 mL/min, as calculated based on CKD-EPI 2021 formula.
* Adequate hepatic function:

  * Total bilirubin ≤ 1.5 × ULN (except for patients with Gilbert's syndrome who are excluded if total bilirubin > 3.0 × ULN or direct bilirubin ≥1.5 × ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 x ULN.
  * Alkaline phosphatase (ALP) ≤ 2.5 x ULN.
* Recovered from any clinically relevant toxicity of the previous chemoradiotherapy cycle unless stable and manageable per investigator´s judgement
* WHO performance status 0-2
* Stable or decreasing corticosteroid dose, or no use of corticoids, for at least 7 days prior to enrollment.
* Baseline brain MRI available, as defined in the schedule of assessments
* Available FFPE tumour tissue from prior neurosurgery for central biobanking and translational research
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within two weeks prior to enrolment.
* Participants of childbearing / reproductive potential should use two adequate methods of birth control, including a highly effective method and a barrier method during the study treatment period and for at least 90 days after the last dose of treatment.

Exclusion Criteria:

* Presence of 1p19q co-deletion, per local assessment.
* Tumour recurrence or progression per RANO 2.0 criteria between first day of radiotherapy and enrolment, per local assessment
* Last chemotherapy dose of first line chemoradiotherapy less than 6 weeks or more than 12 weeks before enrolment
* Prior therapy with an IDH inhibitor or IDH vaccine
* Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Integrated diagnosis of astrocytoma, IDH-mutated, CNS5 WHO grade 4
* Pregnancy or breastfeeding
* Significant known active cardiac disease within 6 months before enrollment, including New York Heart Association Class III or IV congestive heart failure, myocardial infarction, unstable angina, and/or stroke.
* Known hypersensitivity to any of the components of vorasidenib.
* Ongoing use of medications that are CYP2C8, CYP2C9, CYP2C19, or CYP3A substrates with a narrow therapeutic index. Participants must be transferred to other medications before receiving the first dose of study drug.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, known positive human immunodeficiency virus antibody results, or AIDS-related illness.

Participants with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted. Participants with chronic HBV that is adequately suppressed by institutional practice will be permitted.

• Known active inflammatory gastrointestinal disease, chronic diarrhea, previous gastric resection or lap band dysphagia, short-gut syndrome, gastroparesis, or other condition that limits the gastrointestinal absorption of drugs administered orally.

Gastroesophageal reflux disease under medical treatment is allowed (assuming no drug interaction potential).

* Inability or known contraindication to undergo contrast media MRI.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed and discussed with the patient before the enrolment in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2035-04-13 (Estimated); Study Completion 2037-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by local assessment | ~7.7 years and 10.5 years from first patient in
  Progression-free survival (PFS) will be defined as the number of days from date of enrolment to the date of earliest disease progression based on Response Assessment (RANO 2.0) or to the date of death due to any cause, if disease progression did not occur (the date of progression or death or censoring - date of enrolment + 1).
  Patients who received new anti-cancer therapy or cancer-related surgery or radiotherapy prior to progression or death will not be censored at the last assessment where the patient was documented as progression free prior to the new anti-cancer therapy or cancer-related surgery or radiotherapy, instead progression after start of new therapy or surgery will be considered a valid event for PFS.

SECONDARY OUTCOMES:
PFS by local assessment | ~7.7 years and 10.5 years from first patient in
  Progression-free survival (PFS) will be defined as the number of days from date of enrolment to the date of earliest disease progression based on Response Assessment (RANO 2.0) or to the date of death due to any cause, if disease progression did not occur (the date of progression or death or censoring - date of enrolment + 1).
  Patients who received new anti-cancer therapy or cancer-related surgery or radiotherapy prior to progression or death will not be censored at the last assessment where the patient was documented as progression free prior to the new anti-cancer therapy or cancer-related surgery or radiotherapy, instead progression after start of new therapy or surgery will be considered a valid event for PFS.
Progression-free survival (PFS) from the start of radiotherapy | ~7.7 years and 10.5 years from first patient in
  Progression-free survival from the start of radiotherapy will be defined as the number of days from date of start of radiotherapy till progression or censoring with the same rules as for PFS.
Overall Survival | ~7.7 years and 10.5 years from first patient in
  Overall survival (OS) will be defined as the number of days from date of enrolment to the date of death due to any cause (the date of death or censoring - date of enrolment +1). If a subject has not died, the data will be censored at the last date documented to be alive. Patients still alive (or not known to have died before the cutoff date) or lost to follow-up are censored at the last date known to be alive.
Overall Response | ~7.7 years and 10.5 years from first patient in
  All patients included in the study must be assessed for their overall response treatment based on RANO 2.0 criteria at each assessment of the disease, from the start of study treatment until disease progression , even if there is a major protocol treatment deviation, if they are ineligible, or not followed/ /re-evaluated.
  Each patient will be assigned one of the following categories: complete response (CR), partial response (PR), minor response (MR, applicable only to non-enhancing disease), stable disease (SD), Equivocal progressive disease (EqPD), progressive disease (PD), early death (ED) or not evaluable (NE).
  Early death is defined as any death occurring before the first per protocol time point of tumour re-evaluation.
Time to next intervention | ~7.7 years and 10.5 years from first patient in
  Time to next intervention (TTNI) will be defined as the number of days calculated from the date of enrolment until the commencement of further anticancer treatment following vorasidenib or placebo discontinuation (including surgery or radiotherapy), irrespective of whether progression was documented. If a patient does not initiate further anticancer therapy TTNI will be censored at the date of death or last known alive date.
Adverse events | ~7.7 years from first patient in
  All adverse events (AEs) will be recorded; the investigator will assess whether those events are drug related (reasonable possibility, no reasonable possibility) and this assessment will be recorded in the database for all AEs.
  The collection period for all AEs will start up to 4 weeks prior to enrolment and until 30 days after the end of treatment. After those 30 days, only SAEs related to study drug or study participation have to be collected.
  All AEs must be followed until resolution or stabilization.
Health-related Quality of Life QLQ-C30. | ~7.7 years from first patient in
  Health related quality of life (HRQoL) will be measured using a questionnaire which will be completed by the patient: EORTC QLQ-C30
Health-related Quality of Life QLQ-BN20. | ~7.7 years from first patient in
  Health related quality of life (HRQoL) will be measured using a questionnaire which will be completed by the patient: EORTC QLQ-BN20.
Health-related Quality of Life IADL-BN32 | ~7.7 years from first patient in
  Health related quality of life (HRQoL) will be measured using a questionnaire which will be completed by the patient: IADL-BN32
Health-related Quality of Life item list 46 (IL46) | ~7.7 years from first patient in
  Health related quality of life (HRQoL) will be measured using a questionnaire which will be completed by the patient: item list 46 (IL46)
Neurocognitive function HVLT-R - Part A Free recall | ~7.7 years from first patient in
  Neurocognitive function will be measured using a questionnaire which will be completed by the patient: HVLT-R - Part A Free recall
Neurocognitive function TMT - Part A | ~7.7 years from first patient in
  Neurocognitive function will be measured using a questionnaire which will be completed by the patient: TMT - Part A
Neurocognitive function TMT - Part B | ~7.7 years from first patient in
  Neurocognitive function will be measured using a questionnaire which will be completed by the patient: TMT - Part B
Neurocognitive function COWA | ~7.7 years from first patient in
  Neurocognitive function will be measured using a questionnaire which will be completed by the patient: COWA
Neurocognitive function MOS scale | ~7.7 years from first patient in
  Neurocognitive function will be measured using a questionnaire which will be completed by the patient: MOS scale
Neurocognitive function HVLT-R - Part B Delayed recall HVLT-R - Part C Delayed recognition | ~7.7 years from first patient in
  Neurocognitive function will be measured using a questionnaire which will be completed by the patient: HVLT-R - Part B Delayed recall HVLT-R - Part C Delayed recognition
Seizure activity | ~7.7 years from first patient in
  Seizure activity will be measured using will be measured using a questionnaire which will be completed by the physician: Seizure Control Composite Score Index

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Preusser, Study Chair — Universitaetsklinikum Wien - AKH uniklinieken, Vienna, Austria.; Marjolein Geurts, Study Chair — Brain Tumour Center, Erasmus MC Cancer Institute, Rotterdam, the Netherlands.
Locations (33):
- Austria (3):
  - Medical University of Innsbruck, Innsbruck
  - Kepler University Hospital - Neuromed campus, Linz
  - Medical University of Vienna, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - Ghent University Hospital, Ghent
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- Masaryk Memorial Cancer Institute, Brno, Czechia
- France (5):
  - Universitary hospital Bordeaux France, Bordeaux
  - CHU Lyon - Hopital neurologique Pierre Wertheimer, Lyon
  - Marseille APHM, Marseille
  - Assistance Publique Hopitaux de Paris APHP - Sorbonne, Paris
  - Oncopole Claudius Regaud, IUCT-Oncopole, Toulouse
- Germany (5):
  - Universitaskliniken Bonn, Bonn
  - University Hospital Frankfurt -Senckenberg Institute of Neurooncology, Frankfurt
  - NNeurology department heidelberg, Heidelberg
  - Mannheim University Hospital, Mannheim
  - Universitaetsklinikum Regensburg, Regensburg
- Italy (4):
  - Bellaria Hospital, IRCCS Istituto delle Scienze Neurologiche - AUSL di Bologna, Bologna
  - Veneto Institute of Oncology, Padua
  - Sapienza University, Roma
  - AOU Citta della Salute e della Scienza di Torino, Torino
- Netherlands (3):
  - Amsterdam UMC location VUMC, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Erasmus MC, Rotterdam
- Spain (3):
  - Hospital de Sant Pau i La Santa Creu, Barcelona
  - Vall de Hebron Hospital, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Zurich, Zurich
- United Kingdom (4):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - The Christie NHS Foundation Trust, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Royal Marsden Hospital, Surrey Quays